CLINICAL TRIAL: NCT00155194
Title: Impaired T-Lymphocyte Proliferative Function in Biliary Atresia Children With Prolonged Jaundice
Brief Title: Evaluation of Immune Function in Biliary Atresia Children With Prolonged Jaundice
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701170
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-06

CONDITIONS: Biliary Atresia
MeSH Terms: conditions — Biliary Atresia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Null hypothesis of this study: Biliary atresia patients with cholestatic jaundice do not have systemic immunity defect.

DETAILED DESCRIPTION:
Biliary atresia patients with cholestatic jaundice were noted to have increased incidence of infectious complications. Previous animal models of bile duct ligation with acute jaundice ever demonstrated impairment of both humoral and cellular immune function. We performed the immunity study in biliary atresia patients due to the lack of comprehensive systemic immunity study in pediatric cholestatic model. Systemic humoral immunity (total serum IgG, IgA, IgM, C3 and C4), specific cellular immunity (lymphocyte classification, mitogen response, cytokines level after PHA stimulation test), and non-specific cellular immunity (absolute neutrophil count, PMN CD11b/CD18 expression level, PMN superoxide release function, and PMN phagocytosis function) were tested. Association with serum bilirubin level, nutritional status and blood biochemical values were tested to see the relation between systemic immune function and cholestatic jaundice.

ELIGIBILITY:
Inclusion Criteria:

Biliary patients older than 1-year-old status post Kasai operation.

Exclusion Criteria:

Received liver transplantation, immunosuppresant, systemic immunoglobulin (within 6 months) and obvious infectious episode (within 2 weeks).

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2004-04

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Hwei Chang, MD, Study Chair — Department of Pediatrics, Natonal Taiwan University Hospital
Locations (1):
- Department of Pediatrics, National Taiwan University Hospital, Taipei, Taiwan